CLINICAL TRIAL: NCT05351359
Title: mHealth Intervention Delivered in General Practice to Increase Physical Activity and Reduce Sedentary Behaviour of Patients With Prediabetes and Type 2 Diabetes
Brief Title: mHealth Intervention to Increase Physical Activity in Prediabetes and Type 2 Diabetes
Acronym: ENERGISED
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charles University, Czech Republic (Other)
Collaborators: University of Hradec Kralove (Unknown); St George's, University of London (Other); University of Leicester (Other); University Ghent (Other)
Responsible Party: Principal Investigator, Tomáš Větrovský, Lecturer, Charles University, Czech Republic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ENERGISED
Record Dates: First submitted 2022-04-19; First posted 2022-04-28 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-10

CONDITIONS: Type 2 Diabetes; PreDiabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Prediabetic State | interventions — Telemedicine; Crisis Intervention

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active control (Active Comparator): The patients from the active control group will receive brief physical activity advice from their general practitioners at baseline, and they will also receive the Fitbit tracker to self-monitor their daily steps.
  Interventions: Behavioral: Fitbit tracker; Behavioral: brief advice
- Intervention (Experimental): The patients in the intervention group will be exposed to the same procedures as those from the active control group, but will also receive a mHealth-enabled just-in-time adaptive intervention and regular monthly phone counselling in the first 6 months.
  Interventions: Behavioral: mHealth; Behavioral: phone counselling; Behavioral: Fitbit tracker; Behavioral: brief advice

INTERVENTIONS:
Behavioral: mHealth — A mHealth-enabled just-in-time adaptive intervention that is based on the HealthReact system developed by the participating centre at the Faculty of Science of the University of Hradec Kralove. The HealthReact system consists of a server-side application that is connected to the Fitbit server. As such, the system allows for just-in-time text messages triggered by pre-defined context as recorded by the Fitbit wearable monitor. For example, a prompt to take a break from sedentary behaviour can be triggered after 30 sedentary minutes, a suggestion to increase walking cadence can be triggered when continuous, but slow walking is detected, or a motivational message with a specific goal to take more steps to reach their usual daily step count can be triggered when the total daily steps are too low. The mHealth component will be delivered for the entire duration of the study (i.e., 12 months).
  Arms: Intervention
Behavioral: phone counselling — Regular monthly phone calls by trained counsellors support participants in their effort to increase physical activity and reduce sedentary behaviours. The counsellors will use various behaviour change techniques, such as goal-setting, feedback, action planning, etc. The phone counselling will be provided during the first six months, i.e. 6 phone calls will be delivered.
  Arms: Intervention
Behavioral: Fitbit tracker — Fitbit Inspire 2 will be provided by the general practitioner to study participants at the start of the study to enable objective self-monitoring of physical activity.
Behavioral: brief advice — A brief advice will be provided by the general practitioner at the start of the study.

SUMMARY:
Sedentary behaviour has a detrimental effect on the mortality, morbidity, and well-being of patients with type 2 diabetes and prediabetes, and general practitioners should advise patients on how to self-monitor and increase their physical activity. The emergence of mobile health (mHealth) technologies unlocks the potential to further improve physical behaviour using an innovative "just-in-time" adaptive approach whereby behavioural support is provided in real-time, based on data from wearable sensors. Thus, the investigators aim to evaluate the effect of a just-in-time mHealth intervention administered by general practitioners on the physical activity and sedentary behaviour of patients with type 2 diabetes and prediabetes. A total of 340 patients will be recruited from 20 general practices across the Czech Republic and randomly assigned to either an active control or intervention group. Both groups will receive brief physical activity advice from their general practitioners and a Fitbit fitness tracker to self-monitor their daily steps, but the intervention group will also receive a mHealth-enabled just-in-time adaptive intervention and regular monthly phone counselling in the first 6 months. The mHealth intervention will be delivered using a custom-developed system (HealthReact) connected to the Fitbit that will trigger just-in-time text messages. For example, a prompt to take a break from sedentary behaviour will be triggered after 30 sedentary minutes or a motivational message with a specific goal to take more steps will be triggered when the total step count is too low. The primary outcome will be the change in daily step count at 6 months, other outcomes include changes in other physical behaviour measures, blood tests, anthropometry and patient-reported outcomes at 6 and 12 months. If the intervention is effective, this study will provide a model of health prevention that can be directly implemented and commissioned within primary care using existing infrastructure.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of prediabetes or T2DM according to the Czech guidelines for GPs on diabetes mellitus1 and prediabetes2, i.e. fasting plasma glucose 5.6-6.9 mmol/l, or 2-h plasma glucose of 7.8-11.0 mmol/l after ingestion of 75 g of oral glucose load for the diagnosis of prediabetes, and fasting plasma glucose ≥ 7.0 mmol/l, or 2-h plasma glucose ≥ 11.1 mmol/l after ingestion of 75 g of the oral glucose load for the diagnosis of T2DM
* Age 18 years or older.
* Registered at a participating general practice.
* Regular users of a smartphone and willing to use it as part of the study.
* Written informed consent obtained before any assessment related to the study.

Exclusion Criteria:

* unable to walk
* pregnancy
* taking insulin
* living in a residential or nursing care home
* co-morbid conditions that would affect their adherence to the trial procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2022-04-25 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
step count | from baseline to 12-month assessment
  change in daily step count

SECONDARY OUTCOMES:
chair-stand test | at 6 and 12 months
  functional 30s chair-stand test
HbA1c | at 6 and 12 months
  haemoglobin A1c
glycemia | at 6 and 12 months
  fasting plasma glucose
lipid profile | at 12 months
  total cholesterol, LDL cholesterol, HDL cholesterol, triacylglycerids
step count | at 6 months
  change in daily step count
physical behaviour - average acceleration | at 6 and 12 months
  metric of physical activity volume
physical behaviour - intensity gradient | at 6 and 12 months
  metric of physical activity intensity
sedentary time | at 6 and 12 months
  time per day spent sedentary (in minutes)
sedentary bouts | at 6 and 12 months
  time per day (in minutes) spent sedentary in bouts of 30 mins and longer
walking cadence | at 6 and 12 months
  cadence (steps/min) in 5 (non-consecutive) highest-cadence minutes
blood pressure | at 6 and 12 months
  systolic and diastolic blood pressure
Hospital Anxiety and Depression Scale (HADS) | at 6 and 12 months
  symptoms of anxiety and depression: 14 items on a scale 0-3 (a higher score means a worse outcome)
Short Form Survey (SF-12) | at 6 and 12 months
  measure of health-related quality of life: 12 items using various scales converted to a score 0-100 (a higher score means a better outcome)
body mass index | at 6 and 12 months
  weigh in kilograms divided by height in meters squared

CONTACTS AND LOCATIONS:
Overall Officials: Bohumil Seifert, MD, PhD, Study Chair — Charles University, Czech Republic
Locations (1):
- Institute of General Practice, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vetrovsky T, Kral N, Pfeiferova M, Seifert B, Capek V, Jurkova K, Steffl M, Cimler R, Kuhnova J, Harris T, Ussher M, Wahlich C, Malisova K, Pelclova J, Dygryn J, Elavsky S, Maes I, Van Dyck D, Rowlands A, Yates T. mHealth intervention delivered in general practice to increase physical activity and reduce sedentary behaviour of patients with prediabetes and type 2 diabetes (ENERGISED): statistical analysis plan. Trials. 2025 May 20;26(1):166. doi: 10.1186/s13063-025-08865-z. PMID 40394706
- [Derived] Vetrovsky T, Kral N, Pfeiferova M, Kuhnova J, Novak J, Wahlich C, Jaklova A, Jurkova K, Janek M, Omcirk D, Capek V, Maes I, Steffl M, Ussher M, Tufano JJ, Elavsky S, Van Dyck D, Cimler R, Yates T, Harris T, Seifert B. mHealth intervention delivered in general practice to increase physical activity and reduce sedentary behaviour of patients with prediabetes and type 2 diabetes (ENERGISED): rationale and study protocol for a pragmatic randomised controlled trial. BMC Public Health. 2023 Mar 31;23(1):613. doi: 10.1186/s12889-023-15513-1. PMID 36997936